CLINICAL TRIAL: NCT01993641
Title: A Phase II Simon Two-Stage Study of the Addition of Pracinostat to a Hypomethylating Agent (HMA) in Patients With Myelodysplastic Syndrome (MDS) Who Have Failed to Respond or Maintain a Response to the HMA Alone
Brief Title: Phase 2 Study Adding Pracinostat to a Hypomethylating Agent (HMA) in Patients With MDS Who Failed to Respond to Single Agent HMA
Acronym: MEI-005
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Helsinn Healthcare SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEI-005
Record Dates: First submitted 2013-11-14; First posted 2013-11-25 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Myelodysplastic Syndrome; MDS
Keywords: Myelodysplastic Syndrome; MDS; pracinostat; Hypomethylating Agent; HMA; azacitadine; Vidaza; decitabine; dacogen
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — SB939 compound; Azacitidine; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pracinostat added to HMA (Experimental): Pracinostat in combination with HMA treatment (either azacitidine or decitabine) used in initial single agent treatment for that patient
  Interventions: Drug: pracinostat; Drug: Azacitidine; Drug: Decitabine

INTERVENTIONS:
Drug: pracinostat — Histone deacetylase inhibitor (HDACi) Pracinostat is to be taken before HMA administration 3 times/week (e.g., Monday, Wednesday, and Friday) for 3 weeks, followed by 1 week of rest as a 28-day cycle. Pracinostat administration will be at the clinic on Day 1 of Cycles 1 and 2 and subject will self-administer at home on all other days
  Other Names: SB939
Drug: Azacitidine — All patients will receive the dose and schedule of azacitadine to which they previously failed to respond. (e.g. 75 mg/m2 via subcutaneous (SC) injection or intravenous infusion if SC injections are intolerable; 7 days of each 28 day cycle, either Days 1-7, or Days 1-5, rest on Days 6-7, and azacitadine dosing on Days 8-9)
  Other Names: Vidaza
Drug: Decitabine — All patients will receive the dose and schedule of decitabine to which they previously failed to respond. Common 28 day treatment regimens include: 20 mg/m2 IV for either 5 or 10 days of each 28-day cycle, 10 mg/m2 given intravenously daily for first 10 days of each 28 day cycle, or 20 mg/m2 given subcutaneously daily for the first 5 days of each 28 day cycle.
  The 6-week regimen utilizes a dose of 15 mg/m2 by continuous intravenous infusion over 3 hours repeated every 8 hours for 3 days repeated every 6 weeks.
  Other Names: Dacogen

SUMMARY:
The purpose of this open label study is to determine whether combining pracinostat (study drug) with Vidaza (azacitidine) or Dacogen (decitabine) will improve clinical responses in Myelodysplastic Syndrome (MDS) patients who have failed an initial single agent hypomethylating agent (HMA), and to provide additional safety and efficacy data.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent
2. Histologically or cytologically documented diagnosis of MDS (any French-American-British classification [FAB] subtype)
3. Bone marrow blasts >5% and <30% and a peripheral white blood cell (WBC) count of <20,000 /µL
4. Bone marrow biopsy, aspirates, and peripheral blood smears within 28 days of first study treatment
5. Group 1:

   Primary failures: Progression after their most recent HMA therapy according to IWG criteria after receiving single agent azacitidine and/or single agent decitabine, or has worsening cytopenias (increased transfusion requirement), increased BM blasts, progression to a higher FAB type, or develops additional clinically significant cytogenetic abnormalities; Secondary failures: Relapse after any initial CR, PR, HI, or development of clinically significant cytogenetic abnormalities at any time according to IWG criteria after receiving single agent azacitidine or decitabine

   Group 2:

   Failure to achieve a response (any CR, PR or HI) according to IWG criteria definition of stable disease after the most recent HMA therapy (at least 6 cycles of azacitidine or 4 cycles of decitabine)
6. Must have demonstrated tolerability to single agent HMA
7. Able to start combination therapy within 3 months of the last single agent HMA dose with no other therapy for disease under study received during this interval
8. Not a candidate for hematopoietic stem cell transplant within 4 months of screening
9. ECOG performance status of 0, 1, or 2
10. Adequate organ function as evidenced by:

    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x the upper limit of normal (ULN)
    * Total bilirubin ≤1.5 x ULN or total bilirubin of ≤2 mg/dL, whichever is higher
    * Serum creatinine <2 mg/dL, or creatinine clearance ≥60 mL/min
    * QTcF interval ≤470 msec
11. Female or male patients ≥18 years-of-age
12. Male patients with female partners are required to use two forms of acceptable contraception; Female patients of childbearing potential must have a negative pregnancy test ≤7 days before first study treatment.
13. Willingness and ability to understand the nature of this trial and to comply

Exclusion Criteria:

1. Received any of the following within the specified time frame after the last single agent HMA dose until the first administration of study medication:

   * Any therapy for malignancy between the time of single agent HMA and first on-study treatment
   * Hydroxyurea within 48 hours prior to first study treatment
   * Hematopoietic growth factors: erythropoietin, granulocyte colony stimulating factor (G-CSF), granulocyte macrophage colony stimulating factor (GM-CSF), or thrombopoietin receptor agonists within 7 days (14 days for Aranesp) prior to first study treatment
   * Major surgery within 28 days of study day 1
2. Patients who are candidates for aggressive chemotherapy (e.g. typical AML induction therapy)
3. Cardiopulmonary function criteria:

   * Current unstable arrhythmia requiring treatment
   * History of symptomatic congestive heart failure (New York Heart Association Class III or IV)
   * History of myocardial infarction within 6 months of enrollment
   * Current unstable angina
4. Concomitant treatment with agents that have activity against HDAC inhibitors is not permitted
5. Clinical evidence of CNS involvement
6. Patients with gastrointestinal (GI) tract disease, uncontrolled inflammatory GI disease (e.g., Crohn's disease, ulcerative colitis)
7. Active infection with human immunodeficiency virus or chronic hepatitis B or C
8. Life-threatening illness unrelated to cancer or any serious medical or psychiatric illness that could potentially interfere with participation in this study
9. Presence of a malignant disease within the last 12 months, with the exception of adequately treated in-situ carcinomas, basal or squamous cell carcinoma, or non-melanomatous skin cancer and other concurrent malignancies will be considered on a case by case basis
10. Inability or unwillingness (including psychological, familial, sociological, or geographical conditions) to comply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-12; Primary Completion 2015-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Estimate clinical improvement | 6 months
  Clinical Improvement Rate defined as the proportion of patients with CR, Marrow CR, PR, and HI.

SECONDARY OUTCOMES:
Estimate Overall Response Rate (ORR), including all Complete and Partial Responses, Marrow CR, HI, SD, transfusion independence, and cytogenetic responses | 6 months
  Overall Response Rate (ORR), defined as the proportion of patients with CR, PR, Marrow CR, HI, SD, transfusion independence, and cytogenetic responses according to the IWG criteria
Estimate Complete Response (CR) rate | 6 months
  Complete response (CR) rate, defined as the proportion of patients with a confirmed CR (i.e., confirmed by a CBC at least 4 weeks after CR) according to the IWG criteria
Estimate Hematologic Improvement (HI) rate | 6 months
  Hematologic improvement (HI) rate, defined as the proportion of patients who demonstrate major hematologic improvement as defined by the IWG criteria. Only patients with pre-treatment abnormal values will be considered for this endpoint at 8 weeks.
Estimate Duration of Response (DoR) | 6 months
  Duration of Response (for patients who have achieved CR, PR, or HI), defined as the time from the initial determination of response to the time of disease progression or death on study, whichever occurs first. For patients who are alive and have not experienced disease progression on study (prior to receiving subsequent/new treatment or stem cell transplant), duration of response will be censored at the day of the last adequate disease assessment.
Estimate Progression Free Survival (PFS) | 6-12 months
  Progression-Free survival (PFS), defined as the time from first day of study drug administration (Day 1) to either disease progression or death. Patients who have not progressed or are alive will be censored at the date of last adequate disease assessment
Estimate Event Free Survival (EFS) | 12 months
  Event Free Survival (EFS) defined as the time from first day of study drug administration (Day 1) to failure or death from any cause according to the IWG response criteria. Patients who have not progressed, are alive or died without progression will be censored at the date of last adequate disease assessment
Estimate Overall Survival (OS) | 6-24 months
  Overall Survival (OS), defined as the time from the first day of study drug administration (Day 1) to death on study. Patients who are alive will be censored at the date last known alive.
Assess the safety profile of the combination | 12 months
  Assess the adverse event (AE) profile of pracinostat combined with either azacitidine or decitabine by clinical review of safety events by grade, relationship and event outcomes.
Estimate Marrow CR rate | 6 months
  Marrow CR rate, defined as bone marrow <5% myeloblasts and decrease by > 50% over pretreatment according to IWG criteria.
Assess transfusion independence | 6 months
  Transfusion independence, defined as during the treatment period the patient had no RBC transfusions during any 56 consecutive days or more.
Estimate Stable Disease (SD) rate | 6 months
  Stable disease rate defined as failure to achieve at least a PR, but no evidence of progression for > 8 weeks according to IWG criteria.
Estimate Cytogenetic Response rate | 6 months
  Cytogenetic response rate, defined as complete disappearance of the chromosomal abnormality without appearance of new abnormalities, or partial response of at least 50% reduction of the chromosomal abnormality according to IWG criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Garcia-Manero, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (21):
- United States (21):
  - Southern Cancer Center, Mobile, Alabama
  - City of Hope, Duarte, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Sutter Medical Group, Sacramento, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - Florida Cancer Specialist South, Fort Myers, Florida
  - Florida Cancer Specialist North, St. Petersburg, Florida
  - Northwestern University, Chicago, Illinois
  - University of Kansas Cancer Center, Westwood, Kansas
  - University of Kentucky, Lexington, Kentucky
  - John Theurer Cancer Center, Hackensak, New Jersey
  - Oncology Hematology Care, Cincinati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Tennessee Oncology-Chattanooga, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas Southwestern, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Sponsor website — http://MEIPharma.com